CLINICAL TRIAL: NCT06975254
Title: Application and Effect Evaluation of "Internet + Nursing" Scheme Based on Fracture Liaison Service Model in Patients With Hip Fragility Fracture
Brief Title: Application and Effect of "Internet + Nursing" in Hip Fragility Fracture Patients Based on Fracture Liaison Service
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY-2024-241
Record Dates: First submitted 2025-04-02; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Fragility Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Will accept the implementation of the "Internet plus care program" based on the FLS model in additio (Experimental): Informed by previous questionnaire survey results on orthopedic home nursing services-including "Analysis of Current Needs and Influencing Factors for Orthopedic Home Nursing Services" (319 orthopedic patients) and "Survey on Nurses' Willingness and Influencing Factors for 'Internet+ Nursing Services' in Orthopedics" (321 orthopedic nurses)-and through literature review on fracture liaison service (FLS) models, this study employs the Delphi method to develop an FLS-based "Internet+ Nursing" protocol. The protocol focuses on: 1) identifying and intervening in risk factors for recurrent fractures; 2) health education on fall prevention, functional exercise, and osteoporosis management; and 3) delivering continuous post-discharge "Internet+ Nursing" services through multidisciplinary collaboration, including online consultations with orthopedic, rehabilitation, nutrition specialists, and specialized nurses, as well as offline home visits.
  Interventions: Other: On the basis of routine nursing, the "Internet + nursing program" based on the FLS model is implemented
- Will receive routine perioperative care (No Intervention): You will receive routine perioperative care, such as orthopedic doctors and nurses will explain the method, function and significance of early functional exercise by your bed before surgery, and assist in routine functional exercise. After the operation, you will receive routine care, the responsible nurse will evaluate and hand over your situation each shift, and explain the postoperative precautions and rehabilitation exercise methods to you and your family members in the form of IPAD education videos and publicity brochures, and receive a 3-month follow-up

INTERVENTIONS:
Other: On the basis of routine nursing, the "Internet + nursing program" based on the FLS model is implemented — 1) During hospitalization: After the patient is admitted to hospital, the coordinator will establish wechat contact with the patient face to face and establish a good trust relationship with the patient; The coordinator and the doctor will collect the patients' cases together, and then according to the patients' conditions and wishes, the diagnosis and treatment plan will be formulated jointly by multiple disciplines, including medicine, rehabilitation and nutrition management. 2) Before discharge: the coordinator helps the patient to make an appointment for return visit; Issue business cards of the team's online and offline services to patients and guide them to use wechat and online service application procedures (such as Zheli Care and Dr. Nari); 3) After discharge: patients keep in touch with the liaison staff at any time, and any abnormal situation will be contacted by the liaison staff; Team members supervised the patient's medication situation by punching in the mini program
  Arms: Will accept the implementation of the "Internet plus care program" based on the FLS model in additio

SUMMARY:
Fragility fractures, also known as osteoporotic fractures, are fractures that occur as a result of low-energy trauma or minor impact. They are the most serious complication of osteoporosis and are common bone diseases in the elderly. With our country gradually entering the aging society, the incidence of brittle fracture is increasing year by year, most often in the hip. Hip fracture refers to femoral neck, intertrochanteric and subtrochanteric fractures. Due to a series of complications caused by old age, weak body, many underlying diseases, significant decline in self-care ability and other reasons, it is also known as the last fracture in life. According to reports, within 1 year after hip fracture, only 30% of patients can recover to the functional state before fracture, 20% of patients will fracture again, and even cause lifelong disability, seriously affecting the long-term quality of life of patients, the reason may be related to the long course of disease, slow recovery, postoperative nutrition, rehabilitation exercise compliance, self-care ability decline and many other aspects. The fracture liaison service (FLS) is a nurse-centric, multidisciplinary approach to managing osteoporotic fractures that consists of three key elements: The core of identifying patients with fracture risk, assessing fall risk and initiating treatment to prevent refracture is to hire specialized coordinators to link emergency, orthopedics, rehabilitation, nutrition and other departments with community and family services to provide standardized management services for patients, reduce the incidence of refracture and promote the recovery of joint function of patients. Therefore, this study integrates FLS with "Internet + nursing service" and utilizes the advantages of "Internet + nursing service" in informatization to emphasize the risk assessment of re-fracture of patients at home after discharge, home health guidance (such as fall prevention, rehabilitation training and other related knowledge), online consultation of multidisciplinary teams, offline on-site service, etc., so that patients can be discharged from hospital. Access to ongoing medical care reduces the incidence of complications and promotes rapid recovery.

DETAILED DESCRIPTION:
Osteoporotic fractures, also known as fragility fractures, refer to fractures occurring due to low-energy trauma or minor collisions. As the most severe complication of osteoporosis, they are common skeletal diseases in the elderly population . With China's gradual transition into an aging society, the incidence of fragility fractures has increased annually. Hip fractures, the most common type of fragility fracture, involve injuries to the femoral neck, intertrochanteric, and subtrochanteric regions of the femur . Referred to as the "last fracture in life," hip fractures are associated with high morbidity and mortality due to complications arising from advanced age, frailty, multiple comorbidities, and significant declines in self-care ability . Reports indicate that within one year of a hip fracture, only 30% of patients regain their pre-fracture functional status, 20% experience subsequent fractures, and some even face lifelong disability , severely impacting long-term quality of life. These statistics underscore the critical need for standardized management of hip fragility fractures.

Studies have reported that ineffective rehabilitation guidance, insufficient knowledge of rehabilitation training, and lack of scientific self-care capabilities are key factors influencing postoperative recovery in fragility fracture patients . Continuous nursing care, which addresses gaps in in-hospital health education, has become an indispensable component of postoperative care . Since 2015, nursing informatization has been promoted by national policies and plans, emerging as a major trend in nursing development . Driven by rapid technological advancements, the healthcare sector is encouraged to leverage "Internet+ Nursing Services" to explore new models of continuous care . This model, characterized by "online application and offline service," caters to discharged patients or individuals with mobility limitations, meeting their 刚需 for professional nursing services . As a vital component of continuous care, Internet+ Nursing Services play a positive role in rehabilitation guidance and enhancing patient self-management, improving nursing efficiency . However, current challenges exist: most services are provided by part-time clinical nurses without advanced education or referral coordination skills , and physician involvement is limited, leading to incomplete patient assessments during follow-ups. Additionally, reliance on mobile calls and WeChat for follow-ups raises concerns about information reliability. Thus, enhancing the quality of Internet+ Nursing Services for hip fragility fracture patients remains a critical clinical issue.

The fracture liaison service (FLS) is a multidisciplinary management model for osteoporotic fractures , comprising three key elements: identifying patients at fracture risk, assessing fall risk, and initiating treatments to prevent recurrent fractures. Its core involves dedicated coordinators linking emergency, orthopedic, rehabilitation, nutrition, and community services to provide standardized care, reducing fracture recurrence and promoting functional recovery. While FLS has been widely applied in fragility fracture care, its integration with remote nursing remains limited. This study aims to combine FLS with Internet+ Nursing Services, leveraging the informatic advantages of the latter to emphasize post-discharge risk assessment for recurrent fractures, home-based health guidance (e.g., fall prevention, rehabilitation training), online consultations with multidisciplinary teams, and offline home visits. By ensuring continuous medical care after discharge, this integrated model seeks to reduce complications and facilitate rapid recovery.

ELIGIBILITY:
Inclusion Criteria Age ≥ 18 years

Voluntarily signed informed consent

Diagnosis of hip fragility fracture (closed type)

Scheduled for surgical intervention

Adequate communication and comprehension abilities

Ability of patient or caregiver to operate smart electronic devices

Exclusion Criteria History of psychiatric or neurological disorders (e.g., dementia, schizophrenia)

Polytrauma (multiple fractures or major concomitant injuries)

Metastatic cancer, metabolic bone disease, or terminal illness

Insulin-dependent diabetes mellitus

Thyroid disease

Inability to participate due to other medical or social factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily Living Ability Rating Scale (ADL) | 2 weeks, 1 month, 3 months after discharge
  Activities of Daily Living (Barthel Index): Used to assess patients' ability to perform daily living activities. The assessment includes: eating, bathing, grooming, dressing, toileting, mobility, bed-chair transfer, stair climbing, and bowel/bladder control. A total score of 100 indicates complete independence without reliance on others; 61-99 points indicate basic independence in daily life; 41-60 points indicate moderate dependence requiring assistance; 21-40 points indicate significant dependence on others for daily activities; and ≤20 points indicate complete dependence on others.
Harris Hip Joint Function Scale | 2 weeks, 1 month, 3 months after discharge
  Harris Hip Rating Scale: This study uses the Harris Hip Rating Scale, the most widely applied hip assessment tool in North American hip scoring criteria. Developed by Harris in the United States in 1969, the scale consists of 10 items with respective maximum scores as follows: Pain (44 points), Stair climbing (4 points), Putting on and removing shoes and socks (4 points), Sitting in a chair (5 points), Car travel (1 point), Gait (11 points), Walking aid use (11 points), Walking distance (11 points), Deformity (4 points), and Range of motion (5 points). The total score is 100 points, categorized into four grades: excellent (90-100 points), good (80-90 points), fair (70-80 points), and poor (below 70 points).
Complications | 2 weeks, 1 month, 3 months after discharge
  Complications (incidence of recurrent fractures, infection, pressure ulcers, dislocation, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Cheng li Yan, Bachelor, Principal Investigator — The Fourth Affiliated Hospital of Zhejiang UniversitySchool of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No